CLINICAL TRIAL: NCT00991666
Title: Association Between Laser Interferometric Measurement of Fundus Pulsation and Pneumotonometric Measurement of Pulsatile Ocular Blood Flow in Patients With Age-related Macular Degeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. Priv. - Doz. Dr, Medical University of Vienna
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OPHT-200401
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Age-related Macular Degeneration
Keywords: AMD; rigidity; pulsatile ocular blood flow; Physiology of the eye
MeSH Terms: conditions — Macular Degeneration; Muscle Rigidity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): AMD Patients
  Interventions: Procedure: blood flow measurement
- 2 (Active Comparator): healthy controls
  Interventions: Procedure: blood flow measurement

INTERVENTIONS:
Procedure: blood flow measurement — Fundus pulsation amplitude measurement Pulsatile ocular blood flow measurement

SUMMARY:
Several methods have been proposed for the measurement of pulsatile ocular blood flow (POBF). The pneumatic tonometer, which is commercially available, assesses POBF by measurement of intraocular pressure (IOP) changes during the cardiac cycle. The investigators have recently developed a method for the measurement of ocular fundus pulsation, which is based on laser interferometry. In contrast to the Langham system the method is non-contractile and yields a high topographic resolution. Moreover, the pneumatic tonometer assesses the ocular pressure pulse, whereas ocular fundus pulsation is a point measure of the ocular volume pulse. These two parameters are related by the ocular rigidity, which refers to the mechanical properties of the eye coats.

Age-related macular degeneration (AMD) is the most common cause of blindness in the industrialized nations. The mechanisms behind this severe eye disease are, however, still obscure. It has been hypothesized that alterations in choroidal blood flow and ocular rigidity may contribute to the development and progression of AMD. However, there is currently little data to confirm this hypothesis. The present study is an attempt to investigate choroidal blood flow and ocular rigidity by employing laser interferometric measurement of fundus pulsation and pneumotonometric measurement of fundus pulsation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AMD (defined as soft drusen > 63 µm, hyperpigmentation and/or hypopigmentation of the retinal pigment epithelium (RPE), RPE and associated neurosensory detachment, (peri)retinal hemorrhages, geographic atrophy of the RPE, or (peri)retinal fibrous scarring)
* Age between 50 and 90 years

Exclusion Criteria:

* Evidence of any other retinal or choroidal vascular disease
* Regular use of pentoxifylline in the last month before the trial period
* Evidence of a choroidal neovascular membrane
* Diabetes mellitus

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2001-07; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Fundus pulsation amplitude | 10 minutes measurement of FPA
Pulsatile ocular blood flow | 10 minutes measurement of pulsatile ocular blood flow
Ocular rigidity | 10 minutes measurement of ocular rigidity

CONTACTS AND LOCATIONS:
Overall Officials: Leopold Schmetterer, Prof. Dr., Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria